CLINICAL TRIAL: NCT01451723
Title: Phase 2 Randomized Placebo Controlled Trial of Polyphenon E in MS
Brief Title: Safety and Neuroprotective Effects of Polyphenon E in MS; Phase II
Acronym: POEMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unusual high frequency of elevated liver function tests.
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jesus Lovera MD, MD, MsPH, Louisiana State University Health Sciences Center in New Orleans
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23AT004433-02 (NIH); K23AT004433-02 (NIH); K23AT004433 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Polyphenon E; Green tea; EGCG; Epigallocatechin-galleate; Placebo; Randomized controlled trial
MeSH Terms: conditions — Multiple Sclerosis | interventions — polyphenon E; epigallocatechin gallate; Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyphenon E 400mg twice a day (Experimental): Two capsules of Polyphenon E containing 200mg of EGCG each taken twice a day with food.
  Interventions: Drug: Polyphenon E
- Placebo (Placebo Comparator): Matching placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Polyphenon E — Polyphenon E is a standardized green tea extract. For this study we will use capsules of Polyphenon E containing 200 mg of EGCG per capsule. Subjects will take two capsules twice a day with food.
  Other Names: EGCG; epigallocatechin gallate; Green tea extract
  Arms: Polyphenon E 400mg twice a day
Other: Placebo — Matching placebo capsules
  Arms: Placebo

SUMMARY:
The hypothesis is that Polyphenon E can protect brain cells in patients with Multiple Sclerosis. To test this hypothesis we are going to compare the changes in n-Acetyl-Aspartate (a chemical that reflects the number of neurons and their metabolism) over one year between people with MS treated with Polyphenon E at a dose of 400mg twice a day and people with MS treated with a matching sugar pill.

DETAILED DESCRIPTION:
This will be a double blind placebo controlled trial of Polyphenon E as a treatment for MS.

The primary outcome will be the changes in NAA levels over one year. Secondary outcomes will be changes in brain atrophy over one year. As an exploratory outcome we will correlate changes in NAA levels with free Plasma levels of EGCG 8 hours after the morning dose.

Exploratory outcomes include disability progression by EDSS, MS functional composite components and a cognitive test battery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by McDonald criteria
* Relapsing-remitting MS or secondary progressive MS
* Stable therapy with Copaxone, Rebif, Betaseron or Avonex 30 mcg for at least six months
* EDSS Score less than or equal to 7.0
* Ages 18-60.
* Participants must have normal organ and marrow function as defined below:

  1. Leukocytes ≥3,000/µL
  2. Absolute neutrophil count ≥1,500/µL
  3. Platelets ≥100,000/µL
  4. Total bilirubin ≤local upper limit of normal
  5. AST (SGOT) ≤local upper limit of normal
  6. ALT (SGPT) ≤local upper limit of normal
  7. Creatinine ≤local upper limit of normal

Exclusion Criteria:

* MS relapse within the 30 days prior to enrollment
* A primary progressive form of MS.
* Previous treatment prior to study entry as follows: complete radiation ablation of the bone marrow or anti-CD4 antibody treatment (Campath) at any time; mitoxantrone, cyclophosphamide, Natalizumab or other immunomodulatory or immunosuppressant therapies except the DMT's included in the inclusion criteria and methylprednisone for relapses within prior nine months.
* History of renal or liver disease.
* Consumption of green tea or supplements containing green tea or tea extract within 30 days prior to enrollment.
* Participants may not participate in any other clinical trial involving investigational agents during the study, or within six months prior to enrolling in the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Polyphenon E, tea, or any of the inactive ingredients present in the active or placebo capsules, including gelatin.
* History of allergic reactions to gadolinium or any other condition contraindicated for MRI.
* Uncontrolled, clinically-relevant active illness (aside from MS) including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study
* Inability to complete the baseline MRI scan
* Pregnant women
* Any underlying predisposition to gastrointestinal bleeding (peptic ulcer disease, gastritis, diverticulitis, colitis, hemorrhoids)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus F Lovera, MD, Principal Investigator — LSUHSC-New Orleans
Locations (1):
- LSu Health Sciences Center, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Lovera J, Ramos A, Devier D, Garrison V, Kovner B, Reza T, Koop D, Rooney W, Foundas A, Bourdette D. Polyphenon E, non-futile at neuroprotection in multiple sclerosis but unpredictably hepatotoxic: Phase I single group and phase II randomized placebo-controlled studies. J Neurol Sci. 2015 Nov 15;358(1-2):46-52. doi: 10.1016/j.jns.2015.08.006. Epub 2015 Aug 7. PMID 26298797
- See also: LSU MS Clinic — http://www.medschool.lsuhsc.edu/msclinic/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polyphenon E 400mg Twice a Day | Placebo
Started | 6 | 5
Completed | 0 | 0
Not Completed | 6 | 5
Not completed — study halted | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyphenon E 400mg Twice a Day | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (6.2) | 47 (7.6) | 48.2 (6.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in NAA Levels Adjusted for Water Content.
Description: The rate of change will be calculated using all the time points available )baseline, 6 and 12 months) using a mixed model analysis with the Log NAA as the dependent variable and water content, %grey matter, %white matter, %CSF and % lesion volume as covariates. All the voxels available for each subject where estimates have a SD <30 will be used. A spatial anysotropic exponential covariance structure will be used.
Time Frame: 1 year
Population: No subjects completed either the six or twelve month point so no data was available for analysis.
Arm/Group | Polyphenon E 400mg Twice a Day | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Brain Atrophy
Description: Difference between the two groups in brain atrophy as measured by SIENA
Time Frame: 1 year
Arm/Group | Polyphenon E 400mg Twice a Day | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Polyphenon E 400mg Twice a Day | Placebo
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyphenon E 400mg Twice a Day (N=6) | Placebo (N=5)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyphenon E 400mg Twice a Day (N=6) | Placebo (N=5)
elevated liver enzymes (Hepatobiliary disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was halted prematurely because of the high incidence of liver function abnormalities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No